CLINICAL TRIAL: NCT02576002
Title: Study to Estimate the Incidence and Prevalence and Treatment Patterns of Pediatric Pulmonary Hypertension in the US
Brief Title: Epidemiology and Treatment Patterns of Paediatric PAH (Pulmonary Arterial Hypertension)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18515
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric PAH patients: US pediatric population with PAH in MarketScan database during the period 2010-2013
  Interventions: Drug: Assigned pulmonary hypertension medication

INTERVENTIONS:
Drug: Assigned pulmonary hypertension medication — As assigned by treating physician; may include following product classes: - Calcium channel blockers/antagonists - Prostanoids (prostaglandins, thromboxanes, prostacyclines) - Endothelin receptor antagonists - PDE-5 inhibitors - SGc stimulators

SUMMARY:
To describe the prevalence, incidence and current treatment and procedures patterns in a US pediatric population with PAH in MarketScan database during the period 2010-2013

ELIGIBILITY:
Inclusion Criteria:

* All PAH patients who were in the MarketScan database and who were under age 18 at some time during the years 2010 through 2013

Exclusion Criteria:

Not applicable

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will be all patients who were born after 1991 and thus under the age of 18 during the years 2010 to 2013 in the MarketScan data. The larger population of patients under age 18 will comprise the general population from which population-based prevalence rates will be derived.
Sampling Method: Non-Probability Sample
Enrollment: 2691 (Actual)
Dates: Start 2015-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence rate of PAH (pulmonary arterial hypertension) | Retrospective analysis of three year period
Prevalence rate of PAH | Retrospective analysis of three year period

SECONDARY OUTCOMES:
Assigned drug treatment for PAH measured using the MarketScan database | Retrospective analysis of three year period
  Description of pulmonary hypertension-targeted drugs prescribed in the study population and changes during the study period
Diagnostic procedures performed among PAH patients measured using the MarketScan database | Retrospective analysis of three year period
Prevalence of comorbidities among PAH patients | Retrospective analysis of three year period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Boston, Massachusetts, United States